CLINICAL TRIAL: NCT00993070
Title: A Randomized, Crossover, Double Blinded, Placebo Controlled Trial of Topical Capsaicin in Treatment of Painful Diabetic Neuropathy
Brief Title: Efficacy and Safety Study of Topical Capsaicin in Painful Diabetic Neuropathy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Thammasat University (Other)
Collaborators: Bangkok Drug company (Unknown)
Responsible Party: Principal Investigator, Kongkiat Kulkantrakorn, Associate Professor, Thammasat University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MTU-I-1-45/52
Record Dates: First submitted 2009-10-07; First posted 2009-10-09 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Diabetic Polyneuropathy
Keywords: capsaicin; placebo; trial; diabetic polyneuropathy; neuropathic pain
MeSH Terms: conditions — Diabetic Neuropathies; Neuralgia | interventions — Capsaicin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Capsaicin (Experimental)
  Interventions: Drug: Capsaicin
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Capsaicin — 0.025% topical capsaicin applied 4 times per day for 8 weeks
  Other Names: Capsika gel
  Arms: Capsaicin
Drug: placebo — vehicle gel, applied 4 times per day for 8 weeks
  Arms: placebo

SUMMARY:
Painful diabetic neuropathy is the most common cause of neuropathic pain. 0.075% topical capsaicin has been used to treat the pain, but there is no data in lower concentration. This is the efficacy and safety of 0.025% topical capsaicin in treatment of painful diabetic polyneuropathy.

DETAILED DESCRIPTION:
Patient is randomized to receive either 0.025% topical capsaicin or vehicle control (placebo) for 8 weeks. After one week wash-out period, patients will be switched to the other group for 8 weeks.

Outcome will be assessed by visual analog scale, neuropathic pain scale, SF-MPQ, SF-36. Safety and tolerability will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* History of type 2 Diabetes mellitus
* Peripheral neuropathy
* Stabilized on pain medication for at least one month
* No previous invasive intervention for pain relief

Exclusion Criteria:

* Local wound or skin abnormality in the applicable area
* Allergic to capsaicin
* Refuse to participate or give consent
* Has other significant disease or receive medication that may worsen neuropathy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pain relief from pain score reduction, using visual analog scale (VAS) | 8 weeks

SECONDARY OUTCOMES:
Overall clinical improvement, measured by Clinician Global Impression of Change(CGIC) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kongkiat Kulkantrakorn, MD, Principal Investigator — Thammasat University
Locations (1):
- Thammasat University Hospital, Pathum Thani, Thailand